CLINICAL TRIAL: NCT06799078
Title: Racial Disparities in Antidepressant Initiation, Titration, and Adherence After Receiving a Psychiatric Consultation
Brief Title: Racial Disparities in Antidepressant Treatment After a Psychiatric Consultation
Acronym: RITA-PC
Status: Active, not recruiting | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Benoit Mulsant, Senior Scientist, Centre for Addiction and Mental Health
Other Study IDs: 2023-174
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Depression - Major Depressive Disorder; Depression Disorders
Keywords: antidepressant; consultation; depression; major depressive disorder; Race
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants that self-identify as being BIPOC
- Participants that self-identify as being White
  Interventions: Other: Observation while participants receive treatment by their primary care provider

INTERVENTIONS:
Other: Observation while participants receive treatment by their primary care provider — Participants complete a consultation with a psychiatrist who makes some recommendations for the treatment of their depression. The participant's primary care provider decides whether to implement some of these recommendations.
  Groups: Participants that self-identify as being White

SUMMARY:
Patients from black, indigenous, and people of color (BIPOC) communities are reported to have lower rates of antidepressant adherence and response. The investigators have a limited understanding of why this disparity exists. The majority of outpatient psychiatric consultations are one-time assessments that provide treatment recommendations to the primary care provider. It is important to identify whether there are racial differences in accessing and adhering to recommended treatment plans to provide more equitable care. To the investigators' knowledge, there are no studies that examined racial differences in access and barriers to receiving antidepressant treatment after a one-time psychiatric assessment. This study focuses on patients who were diagnosed with major depressive disorder during a psychiatric consultation 3 months prior. We are examining whether there are racial differences in being a) recommended an antidepressant, b) started/switched to a recommended antidepressant, c) treated at a therapeutic dosage, d) adherence to treatment, and e) whether sociodemographic factors, discrimination in medical settings, and patient perception of depression and antidepressant treatment moderate these differences. This study will inform the development of treatment strategies that minimize racial disparities in the treatment of depression.

DETAILED DESCRIPTION:
Overall Design:

The research design of this study combines two online questionnaires, a semi-structured qualitative interview (for a subset of participants), and a structured chart review. All participants who provide consent to participate in the study will be emailed the first online questionnaire a few days later and then the second online questionnaire three months after they have completed their consult. Twenty-four of these participants will also be invited to participate in the semi-structured qualitative interview in addition to the online questionnaires. The participants will have to complete the second online questionnaire prior to the qualitative interview. Chart review will be performed in all participants. Chart review will occur in parallel with the online questionnaires and the interview.

Participants will be recruited from the Centre for Addiction and Mental Health (CAMH) among patients: (1) diagnosed with depression during a one-time psychiatric consultation; (2) who either assent to be contacted regarding potential participation in research during their CAMH consultation, or who have indicated their agreement to be contacted regarding potential participation in research during the CAMH registration process. Potential participants will also be referred to the study by psychiatrists at CAMH after the patient completes a one-time outpatient psychiatric consultation if they assent to be contacted by the research team. Psychiatrists at CAMH will also be provided with REB-approved recruitment pamphlets to give to patients who express an interest in participating in the study, after which the patients can contact the research team directly if they are interested using the contact information provided in the pamphlet.

Shortly after the consultation is completed, potential participants will be contacted to confirm their interest in participation and to obtain informed consent. Shortly after, the participants will be emailed a link to complete a baseline 20-40 minute REDCap online questionnaire. The first online questionnaire will have two parts, the first part including questions about demographic information and the second part including clinical status and previously validated scales. Also, using a structured form adapted from another study conducted at CAMH, the participants' electronic health records will be reviewed to determine the content, structure, and length of the consultation note, the diagnoses given during the consultation, and treatment recommendations, including pharmacological (i.e., names and dosages of psychotropic medications) and non-pharmacological recommendations. Three months after they complete the psychiatric consultation, the participants will be emailed a link to complete the second 10- 20 minute REDCap online questionnaire, assessing treatment processes and outcomes.

In addition, a subgroup of 24 participants will be invited complete a semi-structured qualitative interview after they complete the second survey (using Webex). The participants will have to complete the second online questionnaire prior to the interview. All participants will be invited to take part in both the online questionnaires and the interview at the beginning of the study. This will continue until 12 participants who self-identify as BIPOC and 12 participants who self-identify as White have completed the interview.

Participant Recruitment and Screening:

The target is to have 50 - 100 participants completing the questionnaires, of which half will be participants who self-report as being from BIPOC communities. Invitation to participate in the interview will be offered to all participants from the beginning until 12 participants who self-identify as BIPOC and 12 participants who self-identify as White have completed it.

All potential participants will be contacted by phone by an investigator or a Research Analyst (RA) to screen for eligibility criteria and engage them in a consent discussion.

Sample Size Determination:

Assuming that there will be a 20 - 40% difference between participants who are from BIPOC communities and participants who are White in treatment outcomes (Kales et al., 2013; Simon et al., 2015), α = 0.05, power = 80%, sample size between 46 - 186 participants is sufficient to detect a between-group difference.

A systematic review of qualitative studies reported that the average sample size to reach saturation is 12-13 for homogeneous populations (Hennink & Kaiser, 2022). As the study will consist of at least 2 distinct populations (participants who are White vs. from BIPOC communities), 12 participants from each group is sufficient.

Statistical Methods:

Between-group analyses will be performed by comparing White participants vs. participants from BIPOC communities. If there is a sufficient number of participants from a specific race/ethnicity to perform between-group analyses, secondary analyses will be performed by treating them as a separate group (e.g., White vs. Asian-South vs. Others).

Logistic regression analyses will be used to examine if there is an interaction effect between race/ ethnicity and potential moderators on observed racial disparities in treatment processes. Self-reported gender, annual income, any experience of discrimination in medical settings (DMS scale answer rarely or higher in any of the items), and having a negative perception of antidepressant treatment (Brief IPQ item 4 score < 5) will be explored as potential moderators.

Control of Bias:

Interviewer bias may occur during the semi-structured qualitative interview if the interviewer becomes aware of the participant's race/ ethnicity. To minimize this, interviewers will be unaware of the results of the REDCap questionnaires containing the race/ ethnicity information. Furthermore, interviewers will have a script they have to adhere to.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign and date the informed consent form
2. Stated willingness to comply with all study procedures
3. Age 18 years and older
4. Diagnosis of depression in a psychiatric consultation at CAMH in the last 3 months
5. Not currently followed by a psychiatrist
6. Able to complete the REDCap questionnaire in English using the internet

Exclusion Criteria:

1. Presence of a life-time diagnosis of bipolar disorder or schizophrenia
2. Potential participants with a suicidal plan or intent whose consulting psychiatrist determined are in need of immediate clinical attention (e.g., referral to CAMH ED, voluntary or involuntary hospitalization)
3. Acute psychosis (e.g., MDD with psychotic features)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received an outpatient psychiatric consultation at CAMH within the past 3 months and received a diagnosis of depression, after which they were discharged to the care of their primary care provider
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychotropic medication initiation or change after psychiatric consultation | From the psychiatric consultation to three months after the consultation
  This information will be obtained during the first and second online surveys

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Upon enrolment and 3 months after enrolement
  Measures the severity of depressive symptoms
GAD-7 | Upon enrolment and 3 months after enrolement
  Measures the severity of anxiety symptoms.
Brief Medication Questionnaire (BMQ) | Upon enrolment and 3 months after enrolement
  Used to assess self-reported medication adherence. Also includes a screen for potential nonadherence, belief barriers, and recall barriers to taking the prescribed medication.
Discrimination in Medical Settings scale | Upon enrolment
  Scale for measuring experiences of discrimination in medical settings.
Brief Illness Perception Questionnaire | Upon enrolment
  Measures the patient's perception of consequences of the illness, illness timeline, personal control over their illness, treatment control over their illness, what they view as identifying features of the illness, how much they are concerned about the illness, how well they understand the illness, and their emotional response to their illness
Participant experience during and after their psychiatric consultation. | 3 months after enrolment
  To be captured through a semi-structured qualitative interview which consists of 8-16 open ended questions probing the treatment processes the participants went through after the psychiatric consultation and their experience navigating these processes. The number of questions will depend on their answers. The questions ask the participants to describe their experience of the psychiatric consultation, their understanding and feelings about the diagnosis that was shared with them, what happened after the consultation, what changes (if any) were made to their treatment and why, how they felt about the follow-up appointments (if any) with their family physician, their experience of taking psychotropic medications if any were started or changed, and how they feel about their depression treatment overall.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit H Mulsant, MD, MS, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
This will require additional consent from the study participants as well as REB approval.

REFERENCES:
- [Background] Svarstad BL, Chewning BA, Sleath BL, Claesson C. The Brief Medication Questionnaire: a tool for screening patient adherence and barriers to adherence. Patient Educ Couns. 1999 Jun;37(2):113-24. doi: 10.1016/s0738-3991(98)00107-4. PMID 14528539
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Snowden LR, Thomas K. Medicaid and African American outpatient mental health treatment. Ment Health Serv Res. 2000 Jun;2(2):115-20. doi: 10.1023/a:1010161222515. PMID 11256718
- [Background] Simon GE, Coleman KJ, Waitzfelder BE, Beck A, Rossom RC, Stewart C, Penfold RB. Adjusting Antidepressant Quality Measures for Race and Ethnicity. JAMA Psychiatry. 2015 Oct;72(10):1055-6. doi: 10.1001/jamapsychiatry.2015.1437. No abstract available. PMID 26352783
- [Background] Rossom RC, Shortreed S, Coleman KJ, Beck A, Waitzfelder BE, Stewart C, Ahmedani BK, Zeber JE, Simon GE. ANTIDEPRESSANT ADHERENCE ACROSS DIVERSE POPULATIONS AND HEALTHCARE SETTINGS. Depress Anxiety. 2016 Aug;33(8):765-74. doi: 10.1002/da.22532. Epub 2016 Jun 20. PMID 27320786
- [Background] Peek ME, Nunez-Smith M, Drum M, Lewis TT. Adapting the everyday discrimination scale to medical settings: reliability and validity testing in a sample of African American patients. Ethn Dis. 2011 Autumn;21(4):502-9. PMID 22428358
- [Background] Paradies Y, Ben J, Denson N, Elias A, Priest N, Pieterse A, Gupta A, Kelaher M, Gee G. Racism as a Determinant of Health: A Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 23;10(9):e0138511. doi: 10.1371/journal.pone.0138511. eCollection 2015. PMID 26398658
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kales HC, Nease DE Jr, Sirey JA, Zivin K, Kim HM, Kavanagh J, Lynn S, Chiang C, Neighbors HW, Valenstein M, Blow FC. Racial differences in adherence to antidepressant treatment in later life. Am J Geriatr Psychiatry. 2013 Oct;21(10):999-1009. doi: 10.1016/j.jagp.2013.01.046. Epub 2013 Feb 6. PMID 23602306
- [Background] Ishrat Husain M, Rodie DJ, Perivolaris A, Sanches M, Crawford A, Fitzgibbon KP, Levinson A, Geist R, Kurdyak P, Mitchell B, Oslin D, Sunderji N, Mulsant BH; PARTNERs Study Group. A Collaborative-Care Telephone-Based Intervention for Depression, Anxiety, and at-Risk Drinking in Primary Care: The PARTNERs Randomized Clinical Trial. Can J Psychiatry. 2023 Oct;68(10):732-744. doi: 10.1177/07067437231156243. Epub 2023 Feb 28. PMID 36855791
- [Background] Hennink M, Kaiser BN. Sample sizes for saturation in qualitative research: A systematic review of empirical tests. Soc Sci Med. 2022 Jan;292:114523. doi: 10.1016/j.socscimed.2021.114523. Epub 2021 Nov 2. PMID 34785096
- [Background] Fortuna LR, Alegria M, Gao S. Retention in depression treatment among ethnic and racial minority groups in the United States. Depress Anxiety. 2010 May;27(5):485-94. doi: 10.1002/da.20685. PMID 20336808
- [Background] Donneyong M, Reynolds C, Mischoulon D, Chang G, Luttmann-Gibson H, Bubes V, Guilds M, Manson J, Okereke O. Protocol for studying racial/ethnic disparities in depression care using joint information from participant surveys and administrative claims databases: an observational cohort study. BMJ Open. 2020 Jan 7;10(1):e033173. doi: 10.1136/bmjopen-2019-033173. PMID 31915172
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Breslau J, Cefalu M, Wong EC, Burnam MA, Hunter GP, Florez KR, Collins RL. Racial/ethnic differences in perception of need for mental health treatment in a US national sample. Soc Psychiatry Psychiatr Epidemiol. 2017 Aug;52(8):929-937. doi: 10.1007/s00127-017-1400-2. Epub 2017 May 26. PMID 28550518
- See also: Hayes, A. F. (2022). Introduction to Mediation, Moderation, and Conditional Process Analysis. A Regression-Based Approach (Tgurd ed.). New York: Guilford Press — https://www.guilford.com/books/Introduction-to-Mediation-Moderation-and-Conditional-Process-Analysis/Andrew-Hayes/9781462549030?srsltid=AfmBOoqbNFXLu4YnMqUraR7XMp56CkmEDXiotVfdSXEXZmoJUGxOx1M8
- See also: Rosner, B. (2011). Fundamentals of Biostatistics (7th Ed. ed.): Brooks/Cole. — https://www.unilus.ac.zm/lms/e-books/books/Basic_Sciences/Behavioural%20sciences%20and%20public%20health/Fundamentals%20of%20Biostatistics%20%287th%20Edition%29.pdf